CLINICAL TRIAL: NCT01680406
Title: Ethiopia Antimalarial in Vivo Efficacy Study 2012: Evaluating the Efficacy of Artemether-lumefantrine Alone Compared to Artemether-lumefantrine Plus Primaquine and Chloroquine Alone Compared to Chloroquine Plus Primaquine for Plasmodium Vivax Infection
Brief Title: Ethiopia Antimalarial in Vivo Efficacy Study 2012
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ethiopian Health and Nutrition Research Institute (Other); Federal Minstry of Health of Ethiopia (Other Government); Columbia University (Other); Oromia Regional Health Bureau, Ethiopia (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency); Menzies School of Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-CGH-6338
Record Dates: First submitted 2012-08-30; First posted 2012-09-07 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Plasmodium Vivax Infection
Keywords: Plasmodium vivax; malaria; Ethiopia; Sub-Saharan Africa; primaquine; artemether lumefantrine; chloroquine
MeSH Terms: conditions — Malaria, Vivax; Malaria | interventions — Artemether, Lumefantrine Drug Combination; Primaquine; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Artemether-lumefantrine (Active Comparator): Weight-based dose to be administered as fixed-dose combination twice daily for three days.
  Interventions: Drug: Artemether-lumefantrine combination
- Artemether-lumefantrine and primaquine (Experimental): Artemether-lumefantrine will be given in a weight-based dose to be administered as fixed-dose combination twice daily for three days.
  Primaquine will be given beginning on day 2 of artemether-lumefantrine to patients with a normal G6PD test; dose is weight-based to be administered once daily for 14 days.
  Interventions: Drug: Artemether-lumefantrine combination; Drug: Primaquine
- Chloroquine (Active Comparator): Chloroquine will be given in a weight-based dose to be administered once daily for three days.
  Interventions: Drug: Chloroquine
- Chloroquine and primaquine (Experimental): Chloroquine will be given in a weight-based dose to be administered once daily for three days.
  Primaquine will be given beginning on day 2 of chloroquine to patients with a normal G6PD test; dose is weight-based to be administered once daily for 14 days.
  Interventions: Drug: Primaquine; Drug: Chloroquine

INTERVENTIONS:
Drug: Artemether-lumefantrine combination
  Arms: Artemether-lumefantrine; Artemether-lumefantrine and primaquine
Drug: Primaquine
  Arms: Artemether-lumefantrine and primaquine; Chloroquine and primaquine
Drug: Chloroquine
  Arms: Chloroquine; Chloroquine and primaquine

SUMMARY:
The investigators hypothesize that the addition of primaquine (PQ) to both artemether-lumefantrine (AL) and chloroquine (CQ) for the treatment of Plasmodium vivax infection will result in decreased chance of relapse by about 60%.

The investigators plan to assess the therapeutic efficacy of AL compared to combined AL + PQ and CQ compared to combined CQ + PQ against P. vivax infection. They also plan to determine the number of recurrent vivax episodes in patients receiving PQ compared to those who don't receive PQ. Patients aged above 1 year with symptomatic malaria presenting to health centers will be enrolled for treatment with AL, AL+PQ, CQ, or CQ+PQ for P. vivax infection.

Phase 1 of the study will monitor the clinical, parasitological, and hematological parameters for P. vivax infection over a 42-day follow-up period, which will be used to evaluate drug efficacy. Phase 2 will continue monthly follow-up of these patients for one year to assess frequency of recurring vivax infections. Results from this research study will be used to assist Ethiopia in assessing their current national malaria drug policies.

DETAILED DESCRIPTION:
Following the rapid development of significant drug resistance of Plasmodium falciparum (Pf) to chloroquine and then sulfadoxine-pyrimethamine, artemether- lumefantrine (Coartem or AL) was adopted as first line therapy in Ethiopia in 2004. According to the current national malaria diagnosis and treatment guidelines updated in 2012, first-line treatment for uncomplicated P. falciparum infection is AL. First-line treatment for Plasmodium vivax (Pv) is chloroquine (CQ) alone in malarious areas and with primaquine in non-malarious areas at health center and hospital level. WHO recommends treatment of Pv with CQ or an artemisinin-based combination therapy (ACT) in combination with primaquine. For all clinical infection without laboratory confirmation, AL is the first-line treatment since AL is effective against both Pf and Pv. Thus, in Ethiopia, where treatment for malaria without laboratory confirmation occurs frequently, Pv is often treated with AL as the standard of care. Similarly, the recommended drug for mixed infection with Pf and Pv is AL. Now with wide-spread use of AL and CQ and with evidence that malaria laboratory testing is occurring in about half of those suspected with clinical evidence of malaria infection, the investigators propose to conduct an antimalarial efficacy study to monitor the effectiveness of these therapies in Ethiopia and to determine how efficacious these drugs remain for Pv. In addition, with high rates of relapse with P. vivax infection, the efficacy and safety of co-administering primaquine will be assessed. This information will inform future policy changes with respect to appropriate antimalarial strategies.

ELIGIBILITY:
Inclusion Criteria:

* Slide-confirmed infection with P. vivax
* Age > 1 year
* Lives within 20 km of the enrolling health facility
* Weight ≥ 5.0 kg
* Axillary temperature ≥ 37.5º C or history of fever during the previous 48 hours
* Patient or caregiver agrees to all finger pricks and return visits.

Exclusion Criteria:

* General danger signs or symptoms of severe malaria (see Annex II)
* Signs or symptoms of severe malnutrition, defined as weight-for-age ≤ 3 standard deviations below the mean (NCHS/WHO normalized reference values)
* Slide confirmed infection with any other Plasmodium species. besides P. vivax mono-infection
* Acute anemia, defined as Hg < 8 g/dl
* Known hypersensitivity to any of the drugs being evaluated
* Presence of febrile conditions caused by diseases other than malaria
* Serious or chronic medical condition by history (cardiac, renal, hepatic diseases, sickle cell disease, HIV/AIDS)
* Pregnant or breastfeeding women.
* History or hemolysis or severe anemia
* Regular medication, which may interfere with antimalarial pharmacokinetics

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
P. vivax treatment failures following treatment with AL compared to AL+PQ | day 28 and 42
P. vivax treatment failures following treatment with CQ compared to CQ+PQ | day 28 and 42

SECONDARY OUTCOMES:
Number of episodes of P. vivax parasitemia over one year following initial effective therapy against P. vivax (i.e. parasite clearance) | 1 year after day 0 of enrollment

OTHER OUTCOMES:
Safety endpoint | baseline (day 0) and day 28
  Change in hemoglobin concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jimee Hwang, MD MPH, Principal Investigator — Centers for Disease Control and Prevention; Tesfay Abreha, MSc, MPH, Principal Investigator — ICAP-Columbia University, Addis Ababa, Ethiopia; David Hoos, MD MPH, Principal Investigator — ICAP-Columbia University, New York, USA
Locations (2):
- Ethiopia (2):
  - Bishoftu Malaria Center, Bishoftu
  - Batu Health Center, Zeway

REFERENCES:
- [Derived] Kleinecke M, Sutanto E, Rumaseb A, Hoon KS, Trimarsanto H, Osborne A, Manrique P, Peters T, Hawkes D, Benavente ED, Whitton G, Siegel SV, Pearson RD, Amato R, Rai A, Nhien NTT, Nguyen HC, Assefa A, Degaga TS, Abate DT, Rahim AG, Pasaribu AP, Sutanto I, Alam MS, Pava Z, Lopera-Mesa T, Echeverry D, William T, Anstey NM, Grigg MJ, Day NP, White NJ, Kwiatkowski DP, Taylor AR, Noviyanti R, Neafsey D, Price RN, Auburn S. Microhaplotype deep sequencing assays to capture Plasmodium vivax infection lineages. Nat Commun. 2025 Aug 5;16(1):7192. doi: 10.1038/s41467-025-62357-x. PMID 40764298
- [Derived] Abreha T, Hwang J, Thriemer K, Tadesse Y, Girma S, Melaku Z, Assef A, Kassa M, Chatfield MD, Landman KZ, Chenet SM, Lucchi NW, Udhayakumar V, Zhou Z, Shi YP, Kachur SP, Jima D, Kebede A, Solomon H, Mekasha A, Alemayehu BH, Malone JL, Dissanayake G, Teka H, Auburn S, von Seidlein L, Price RN. Comparison of artemether-lumefantrine and chloroquine with and without primaquine for the treatment of Plasmodium vivax infection in Ethiopia: A randomized controlled trial. PLoS Med. 2017 May 16;14(5):e1002299. doi: 10.1371/journal.pmed.1002299. eCollection 2017 May. PMID 28510573